CLINICAL TRIAL: NCT02301455
Title: REACH OUT: to Reduce High Blood Pressure in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lesli E. Skolarus, MD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00091668
Record Dates: First submitted 2014-10-23; First posted 2014-11-26 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Hypertension; Stroke
Keywords: hypertension treatment; stroke prevention
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control, Not hypertensive (No Intervention): Participants who after 3 weeks do not have high blood pressure or are not responsive to text messages.
- Text messages, hypertensive (Experimental): Participants who after 3 weeks have high blood pressure and are responsive to text messages, who are then randomized to receive text messages.
  Interventions: Behavioral: Text messaging
- No text messages, hypertensive (No Intervention): Participants who after 3 weeks have high blood pressure and are responsive to text messages, who are then randomized to not receive text messages.

INTERVENTIONS:
Behavioral: Text messaging — persistently hypertensive participants will be randomized to receive these tailored, motivational text messages
  Arms: Text messages, hypertensive

SUMMARY:
One of the most powerful predictors of stroke is hypertension, with estimates of approximately 33% of adults in the United States experiencing this condition.

Hypertension is very prevalent in the emergency department (ED), but significantly undertreated. The overall goal of this project is to develop a text messaging intervention to improve hypertension care in the ED. This will first be done by testing the feasibility of identifying hypertensive patients in the ED, and the response rate to text messages.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 y/o)
* At least one BP of systolic blood pressure (SBP) ≥160 or a diastolic blood pressure (DBP) ≥100 or only BP performed prior to enrollment is SBP ≥160 or a DBP ≥100 (If the patient has repeated measurements after achieving Criteria 1, but prior to being enrolled, at least one of the repeat BP remains SBP ≥140 or a DBP ≥90)
* Must have mobile phones with text-messaging capability
* Likely to be discharged from the ED

Exclusion Criteria:

* Adult who is in an urgent condition
* Unable to read
* Non-English speaking
* Incarcerated/ institutionalized resident
* Pregnant, or has a pre-existing condition that makes follow-up for 4 months unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of people who respond to text messages and are persistently hypertensive | 3 weeks

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure | 4 months
Feasibility of a screening algorithm | 4 months
  Proportion of subjects recruited compared to proportion of subjects approached. Subject eligibility identified by screening algorithm.
Feasibility of subject follow-up mechanism | 4 months
  Proportion of subjects responding to follow-up text messages
Mean group differences and standard deviations for systolic blood pressure | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Meurer WJ, Dome M, Brown D, Delemos D, Oska S, Gorom V, Skolarus L. Feasibility of Emergency Department-initiated, Mobile Health Blood Pressure Intervention: An Exploratory, Randomized Clinical Trial. Acad Emerg Med. 2019 May;26(5):517-527. doi: 10.1111/acem.13691. Epub 2019 Feb 19. PMID 30659702